CLINICAL TRIAL: NCT01548469
Title: Single Blind, Randomized, Active-controlled Comparative Clinical Trial to Evaluate Clinical Efficacy and Safety Following the Application for 4 Weeks of Bio Mineral Toothpaste in Patients With Mild Periodontitis
Brief Title: Study to Evaluate Clinical Efficacy and Safety of Bio Mineral Toothpaste in Patients With Mild Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Youngkyung Ko, Assistant professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIRUS_DENTAL
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Periodontitis
Keywords: Mild periodontitis; Bio Mineral toothpaste; Geumjin Thermal Water
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perio Total Care toothpaste (Active Comparator): A Group which use Perio Total Care toothpaste during participation.
  Interventions: Other: Perio Total Care toothpaste
- Bio Mineral toothpaste (Experimental): A Group which use Bio Mineral toothpaste during participation.
  Interventions: Other: Bio Mineral toothpaste

INTERVENTIONS:
Other: Bio Mineral toothpaste — Frequency: 2 times everyday/Duration: 4 weeks/Dosage: 1ml at once
  Arms: Bio Mineral toothpaste
Other: Perio Total Care toothpaste — Frequency: 2 times everyday/Duration: 4 weeks/Dosage: 1ml at once
  Arms: Perio Total Care toothpaste

SUMMARY:
The hypothesis of this study is that using "Bio Mineral" toothpaste for 4 weeks will decrease plaque and gingivitis of mild periodontitis patients compared to patients using "Perio Total Care" toothpaste.

This study is Single blind, Randomized, Active-controlled Comparative clinical trial to evaluate clinical efficacy and safety following the application for 4 weeks of Bio Mineral toothpaste in patients with mild periodontitis.

DETAILED DESCRIPTION:
This study is Single blind, Randomized, Active-controlled Comparative clinical trial to evaluate clinical efficacy and safety following the application for 4 weeks of Bio Mineral toothpaste in patients with mild periodontitis. 30 patients of treatment group and 30 patients of control group, total 60 patients will be enrolled to this study. Every patients will use investigational toothpaste 2 times everyday for 4 weeks and brush their teeth at least 3 minutes each time with 1ml of toothpaste.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy man or menopausal woman who is at least 18 to maximum 63 years of age.
2. Agreed to participate voluntarily in the study.
3. Must have over 20 maxillary teeth
4. Must have mild periodontal disease which can induce mild plaque.
5. Having no general disease except for dental disease.
6. Must be able to understand and carry out the trial's objective and method.

Exclusion Criteria:

1. Who has history of using antimicrobials or antibiotics during the past 30 days.
2. Who has history of periodontal treatment during the past 30 days.
3. Who has acute pain or severe suppuration caused by pericoronitis of the wisdom tooth.
4. Who has hypersensitive conditions caused by Gingivitis or periodontitis.
5. Who having restorative dentistry or wearing braces widely.
6. Who using tobacco products (Except for who quit smoking)
7. Who has been participated in other clinical trials during the past 4 weeks.
8. Who judged inappropriate to participate in the study by investigator

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Changes in score of "Turesky Modification of the Quigley-Hein Plaque Index" at 4 weeks from baseline. | 0 to 4 weeks
  Changes in score of "Turesky Modification of the Quigley-Hein Plaque Index" at 4 weeks from baseline.
Changes in score of "Modified Gingival Index" at 4 weeks from baseline. | 0 to 4 weeks
  Changes in score of "Modified Gingival Index" at 4 weeks from baseline.

SECONDARY OUTCOMES:
Changes in score of "BOP(Bleeding on probing)" at 4 weeks from baseline. | 0 to 4 weeks
  Changes in score of "BOP(Bleeding on probing)" at 4 weeks from baseline.
Compare Satisfaction of treatment group to Control Group at 4 weeks using Satisfaction Questionnaire. | 4 weeks
  Compare Satisfaction of treatment group with Control Group at 4 weeks using Satisfaction Questionnaire.
  Questionnaire Item
  1. Elimination of plaque
  2. Feeling of refreshment
  3. Amount of bubble.
  4. Feeling of flow.
  5. Taste and Flavor.
  6. Level of cleansing teeth
  7. Creamy consistency
  Each subjects will rate score 0(Very dissatisfied) to 10(Very satisfied) using VAS(Visual Analog Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Youngkyung Ko, M.D., Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seocho-Gu, Seoul, South Korea